CLINICAL TRIAL: NCT01504828
Title: Cardiac Energetics and Function in Normal Human Ageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BH111454; 95309 (Other: Northumberland Tyne and Wear CLRN)
Record Dates: First submitted 2011-12-21; First posted 2012-01-05 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Left Ventricular Function Systolic Dysfunction; Left Ventricular Function Diastolic Dysfunction; Ageing
Keywords: Energy Metabolism; Ageing; left ventricle; energetics; function
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramipril (Experimental): Those who are 40 years and older receive an ACE inhibitor to determine if this reduces age-related changes in left ventricular energetics and function
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — Ramipril in one dose to reduce vascular stiffness to determine effects of this on left ventricular function and energetics

SUMMARY:
Normal aging is characterized by altered cardiovascular function. Our preliminary data with MR imaging and spectroscopy in normal subjects without cardiovascular disease or hypertension show that age-related cardiac dysfunction is characterized initially by impaired relaxation of the heart (40 - 60 years), and then at > 60 years altered contraction and impaired myocardial energetics. For the first time, the investigators will test whether the functional and energetic effects of normal aging can be reversed by acutely reducing stiffness of peripheral blood vessels using an ACE inhibitor. This will potentially have important insights into how normal aging affects the heart, and how potential treatments could be used to attenuate this process.

DETAILED DESCRIPTION:
Normal aging is characterized by altered cardiovascular function. Our preliminary data with MR imaging and spectroscopy in normal subjects without cardiovascular disease or hypertension show that age-related cardiac dysfunction is characterized initially by diastolic dysfunction (40 - 60 years), and then at > 60 years altered systolic strains and impaired myocardial energetics. The investigators propose to study the mechanism of these findings in subjects with normal aging without any cardiovascular disease, hypothesizing that increased vascular stiffening contributes to impaired energetics and left ventricular function. For the first time, the investigators will test whether the functional and energetic effects of normal aging can be reversed by acutely reducing afterload using an ACE inhibitor. This will be tested at 2 ages (40-60 and > 60 years), so that the intervention tests the hypothesis soon after the abnormalities develop (40-60 years - diastolic dysfunction; > 60 years energetics and altered strains). This will potentially have important insights into how normal aging affects the heart, and how potential treatments could be used to attenuate this process.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 20 and 80 years

Exclusion Criteria:

* Any cardiovascular condition including hypertension, or on any cardiovascular therapy.
* Blood Pressure > 150 mmHg systolic, and/or > 90 mmHg diastolic
* Claustrophobia
* Implanted metal prosthesis
* Chronic renal failure requiring dialysis
* Diabetes mellitus.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Vascular Stiffness | 2 Hours - Acute study with no follow-up
  There are 3 principal measures of vascular stiffness, and these are central pulse pressure, central systolic pressure, and the augmentation index. These are correlated against the 3 principal measures of left ventricular function and energetics that are known to change with age: torsion to shortening ratio, early to late diastolic filling ratio, and the ratio of phosphocreatine to adenosine triphosphate (listed as separate Primary Outcome Measures).
Left Ventricular Energetics | 2 hours - Acute Study, no follow-up
  Left ventricular energetics is measured as the ratio of phosphocreatine to adenosine triphosphate
Left Ventricular Function | 2 hours - Acute Study, no follow-up
  Left ventricular function is measured with the 2 parameters that are known to change with age: ratio of early to late diastolic filling, and ratio of torsion to shortening ratio.

SECONDARY OUTCOMES:
Effects of ACE inhibitor on left ventricular energetics and function in those subjects aged 40 and over | 6 hours - Acute study, no follow-up
  A single dose of ACE inhibitor is given to reduce vascular stiffness, and we then measure the effects of this on the measures of left ventricular function and energetics which are the torsion to shortening ratio, diastolic early to late filling ratio, and the phosphocreatine to adenosine triphosphate ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Guy A MacGowan, MD, Principal Investigator — Freeman Hospital, Newcastle upon Tyne and Newcastle University
Locations (1):
- Campus for Ageing and Vitality, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Hollingsworth KG, Blamire AM, Keavney BD, Macgowan GA. Left ventricular torsion, energetics, and diastolic function in normal human aging. Am J Physiol Heart Circ Physiol. 2012 Feb 15;302(4):H885-92. doi: 10.1152/ajpheart.00985.2011. Epub 2011 Dec 16. PMID 22180656
- [Derived] Parikh JD, Hollingsworth KG, Kunadian V, Blamire A, MacGowan GA. Measurement of pulse wave velocity in normal ageing: comparison of Vicorder and magnetic resonance phase contrast imaging. BMC Cardiovasc Disord. 2016 Feb 19;16:50. doi: 10.1186/s12872-016-0224-4. PMID 26892669